CLINICAL TRIAL: NCT00849927
Title: Circumferential Lesions of the Glenoid Labrum: A Prospective Cohort Study of Arthroscopic Repair With Minimum 2-Year Follow-up: A Multi-Center Study.
Brief Title: Circumferential Lesions of the Glenoid Labrum
Status: Completed | Type: Observational
Sponsor: Society of Military Orthopedic Surgeons (Network)
Responsible Party: John M. Tokish, Chief Sports Medicine, USAF Academy, Society of Military Orthopedic Surgeons
Other Study IDs: somos 12-04-01
Record Dates: First submitted 2009-02-18; First posted 2009-02-24 (Estimated); Last update posted 2009-02-24 (Estimated); Status verified 2009-02

CONDITIONS: Shoulder Instability
Keywords: shoulder instability; labral lesions; arthroscopic labral repair; SLAP; triple labrum; circumferential labrum; Pan-labral lesion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Objective: Symptomatic pan-labral or circumferential (360 degree) tears of the glenohumeral labrum are an uncommon injury. The purpose of this study is to report the prospective surgical results of circumferential lesions of the glenoid labrum using validated outcome instruments.

Methods: From July 2003 to May 2006, 41 shoulders in 39 patients with mean age of 25.1 years (range, 17 to 38) were prospectively enrolled in a multi-center study (3 surgeons) and treated for a circumferential (360-degree) lesion of the glenoid labrum. There were 34 men and 5 women, all with a primary diagnosis of pain and recurrent shoulder instability. All patients underwent arthroscopic repair of the circumferential labral tear with a mean of 7.1 suture anchors (range, 6 to 9). The outcomes in 39 of 41 shoulders (92.7% follow-up) were assessed at a mean final follow-up of 31.8 months (range, 24 to 53 months) with VAS pain and instability scales (0 to 10), a physical examination, the Single Assessment Numeric Evaluation Score (SANE), the American Shoulder and Elbow Surgeons Score (ASES), and the SF-12 score.

DETAILED DESCRIPTION:
Patient Demographics A total of 41 shoulders (34 men, 5 women) with mean age of 25.1 years (range, 17 to 38 years) were prospectively enrolled. The outcomes in 39 of 41 shoulders (92.7% follow-up) were assessed at a mean final follow-up of 31.8 months (range, 24 to 53 months). Thirty-seven of 39 patients were right handed. The dominant shoulder was affected in 30 shoulders, non-dominant in 11. Every patient had a primary chief complaint of shoulder pain with a history of anterior and/or posterior shoulder instability. All had a traumatic onset of their symptoms, twelve as a result of contact sports and had failed initial non-operative management. Two patients had had a previous operation, including one patient with a previous open Bankart, 4 years prior to index operation, and another that had a previous posterior arthroscopic "labral repair" which subsequently sustained an anterior dislocation. This was revised with open inferior capsular shift, 2 years prior to index operation. Twenty-six shoulders presented with clear evidence of primary anterior instability. These patients clearly remembered the initial dislocation event and demonstrating an abducted-externally rotated arm at the time of dislocation. Twenty-four of these patients also had pre-reduction radiographs showing anterior dislocation. An additional five patients in the group had variable levels of glenoid bone loss (5-10%), with small Hill-Sachs injuries. Nine shoulders had clear evidence of posterior instability as evidenced by these patients clearly remembering their initial dislocation event, and demonstrating a forward flexed, adducted, and internally rotated position of the arm at the time of dislocation. The remaining six shoulders could not discern between anterior or posterior instability as a primary direction.

All physical examinations were performed by the treating orthopedic surgeon. All shoulders were compared to the contralateral side for range of motion, strength, tenderness, and provocative maneuvers. Range of motion was examined in forward flexion, abduction, and external and internal rotation at 00 and 90 0 of abduction. As part of our normal protocol, values not significantly different from the contralateral side were recorded as "normal". Any value noted to be abnormal was to be recorded in degrees, or in the case of internal rotation at 00, the spinal level. On physical examination no patient was noted to have a significant loss of active or passive motion in flexion, abduction, internal rotation, or external rotation at 00. Thirty-nine of the 41 shoulders demonstrated a positive apprehension sign20, and thus arms were not taken to maximum external rotation in the abducted position in these patients. Strength testing was accomplished with manual muscle testing compared to the opposite arm in all 39 patients. Specific testing included shoulder abduction, internal and external rotation at 00, resisted scaption, lift-off and belly press testing20, as well as elbow flexion and extension, wrist flexion and extension, and interosseous muscle testing. No significant deficit was noted in any of these positions. All patients had pain induced limitation of strength testing during an active compression test20. Provocative maneuvers included anterior and posterior load and shift testing, an anterior apprehension test, a push-pull test for posterior instability, and an active compression test20 . Thirty-nine of 41 shoulders had a positive apprehension test20. Care was taken to place the patient with their arm in 90 degrees of abduction and increasing external rotation. Patients were asked to discern when they became symptomatic, and then asked whether the shoulder felt like it was "coming out" or if their symptoms were just pain. A positive apprehension test was defined as a sensation of the former. All 39 patients had a positive push-pull test for posterior laxity 20and pain. This test is performed by placing the patient supine on the examining table with the arm placed in 90 degrees of abduction and neutral rotation. The wrist is grasped and "pulled" by the examiner with one hand, while the other hand is used to "push" the shoulder backward. A positive test is signified by subluxation of the joint with a reproduction of the patient's symptoms. Impingement signs including Neer's sign, Hawkin's sign, and painful arc were performed on all 39 patients 20. At least one of the signs was positive in all patients. An active compression test was performed on all 39 patients, and noted to be positive with pain and weakness in all patients. No patient demonstrated an increased sulcus sign, or any sign of hyperlaxity.

MRIs were obtained in all 41 shoulders and all radiologic reports were reviewed. Thirty of 41 of these MRI's were done in conjunction with a gadolinium contrast arthrogram. Intraoperatively, all patients underwent an examination under anesthesia with particular attention directed toward anterior and posterior laxity examinations compared to the opposite side according to the grading system for instability established by the American Shoulder and Elbow Surgeons 21,22. Inferior laxity was measured by a sulcus sign measured in centimeters from the edge of the acromion to the top of the humeral head. At arthroscopy, all patients demonstrated complete circumferential tear of the glenoid labrum. One patient had an additional complete radial split of the labrum at the 1 o'clock position (anteriorly), which was repaired. The average patient had 7.1 anchors placed (range, 6-9). Post-operative examination while still under anesthesia showed restoration of normal anterior and posterior glenohumeral translation "to the rim".

Post-operatively, patients were seen at 2 weeks, 6 weeks, and 3 months, 6 months, one year, and yearly after that. History was taken with particular attention to recurrence of dislocation or feelings of apprehension or pain. Physical examination beginning at 3 months assessed range of motion, anterior apprehension, and posterior reproduction of symptoms using a push-pull test20. In addition, strength testing was accomplished, as was an active compression test. Patient outcomes were re-accomplished for the SANE, modified ASES and SF-12 visits at each follow-up visit beginning at 6 weeks. In addition, each patient was asked if he or she would undergo the surgery again. All surveys were administered using a standard form, and entered into the SOMOS database. Data was combined among surgeons using de-identified patient data.

ELIGIBILITY:
Inclusion Criteria:

* Surgical documentation of Pan Labral Lesion of shoulder
* Pre-operative documentation of outcomes scores

Exclusion Criteria:

* lacking a Pan labral lesion
* other confounding pathology such as nerve deficit, chondral damage, rotator cuff tear

Ages: 17 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Department of Defense active duty members
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2003-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
ASES score | 5 years

SECONDARY OUTCOMES:
VAS pain | 5 yrs
Visual Analog Score Instability | 5 years
SANE score | 5 yrs
SF-12 score | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: John M Tokish, MD, Principal Investigator — Society of Military Orthopedic Surgeons
Locations (2):
- United States (2):
  - Navy Medical Center San Diego, San Diego, California
  - US Air Force Academy, Colorado Springs, Colorado

REFERENCES:
- [Result] Lo IK, Burkhart SS. Triple labral lesions: pathology and surgical repair technique-report of seven cases. Arthroscopy. 2005 Feb;21(2):186-93. doi: 10.1016/j.arthro.2004.09.022. PMID 15689868